CLINICAL TRIAL: NCT02689245
Title: Randomized Controlled Trial Comparing the Efficacy and Safety of FMT in Hepatitis B Reactivation Leads to Acute on Chronic Liver Failure.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-ACLF-007
Record Dates: First submitted 2016-02-13; First posted 2016-02-23 (Estimated); Last update posted 2018-11-23 (Actual); Status verified 2018-02

CONDITIONS: Acute on Chronic Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure | interventions — Tenofovir; Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tenofovir + Fecal Microbiota Transplantation (FMT) (Experimental)
  Interventions: Drug: Tenofovir; Drug: Fecal Microbiota Transplantation (FMT)
- Tenofovir (Active Comparator)
  Interventions: Drug: Tenofovir

INTERVENTIONS:
Drug: Tenofovir
Drug: Fecal Microbiota Transplantation (FMT)
  Arms: Tenofovir + Fecal Microbiota Transplantation (FMT)

SUMMARY:
Data for stool microbiome will be collected for all the chronic hepatitis B subjects (pre cirrhotic,compensated,decompensated and reactivation). All the in and out patient with Hepatitis B reactivation will be recruited and randomized into two arms.

Group 1 Tenofovir Group 2 Tenofovir with FMT (Fecal Microbiota Transplant).

Tenofovir would be given 300 mg once daily FMT through NJ (Naso-Jejunal) tube for 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. Reactivation of Chronic Hepatitis B Virus leads to Acute on Chronic Liver Failure- (MELD (Model for End Stage liver Disease) >18 years.
2. 18-75 yr both male and female
3. Chronic Hepatitis B patient (precirrhotic,compensated,decompensated).
4. Healthy adult family member of the patient will be taken as a control.

Exclusion Criteria:

* Acute on Chronic Liver Failure due to other causes -Alcohol,Hepatitis A Virus,Hepatitis E Virus,HSV (Herpes Simplex Virus),CMV (Cytomegalovirus),EBV (Epstein-Barr Virus) other hepatotropic virus,Drugs,CAM.
* Active gastrointestinal bleeding
* Intracranial bleeding
* Multi-organ failure (>2) on mechanical ventilation
* SOFA score >2
* On high inotropic support
* Paralytic ileus
* Pregnancy
* Hepatocellular Carcinoma
* Antibiotic,probiotic within last 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-02-26 (Actual); Primary Completion 2018-03-13 (Actual); Study Completion 2018-03-13 (Actual)

PRIMARY OUTCOMES:
Transplant free survival. | 3 months

SECONDARY OUTCOMES:
Reduction in Hepatitis B Virus DNA level ≥ 2 log. | 2 weeks
Improvement in MELD (Model for End Stage Liver Disease) score. | 2 weeks
Improvement in CTP (Child Pugh Turcotte) score. | 2 weeks
Mortality | 1 Month
Mortality | 3 Months
Improvement in hepatic Encephalopathy. | 7 days
  Improvement is defined as reduction in grading (severity) of hepatic encephalopathy from baseline value.
Improvement in International Normalized ratio. | 7 days
  Improvement is defined as International Normalized ratio value within normal limits
Improvement in Total bilirubin. | 7 days
  Improvement is defined as Total bilirubin value within normal limits.
Development of infectious complications during follow up in both groups | 7,15,30 and 90 days
Improvement in APACHE (Acute Physiology and Chronic Health Evaluation) score in both groups | 7,15,30 and 90 days
Improvement in SOFA (Sequential organ failure assessment) score in both groups. | 7,15,30 and 90 days
Change in gut microbiome in both the groups | 0,7,15,30 and 90 days
Assessment of organ failures in both groups | 7,15,30 and 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Dr Juned Ahmad, MD, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided